CLINICAL TRIAL: NCT03631511
Title: Histological Evaluation of Direct Pulp Capping on Human Pulp Tissue Using a RetroMTA
Brief Title: Histological Evaluation of Hard Tissue Formation After Direct Pulp Capping With RetroMTA
Acronym: RetroMTA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pomeranian Medical University Szczecin (Other)
Responsible Party: Principal Investigator, Alicja Nowicka, DDS, PhD Alicja Nowicka, Pomeranian Medical University Szczecin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Direct capping RetroMTA
Record Dates: First submitted 2018-07-24; First posted 2018-08-15 (Actual); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Dental Pulp Exposure
Keywords: direct pulp capping, RetroMTA, histological evaluation
MeSH Terms: conditions — Dental Pulp Exposure | interventions — mineral trioxide aggregate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RetroMTA (Experimental): Direct pulp capping with RetroMTA (BioMTA, Daejeon, Korea)
  Interventions: Procedure: direct pulp capping with RetroMTA

INTERVENTIONS:
Procedure: direct pulp capping with RetroMTA — The study included seven caries-free third molars from three adults. These teeth were subjected to pulp exposure, direct capping with RetroMTA, and restoration with a composite resin. Seven months later, the teeth were clinically and radiographically evaluated. The teeth were then extracted and subjected to histological processing and evaluation.

SUMMARY:
This study presents a clinical and histological evaluation of human pulp tissue responses after direct capping using RetroMTA. Seven teeth were subjected to pulp exposure, direct capping with RetroMTA, and restoration with a composite resin. Seven months later, the teeth were clinically and radiographically evaluated. The teeth were then extracted and subjected to histological processing and evaluation.

DETAILED DESCRIPTION:
The study was conducted in accordance with the tenets of the World Medical Association Declaration of Helsinki. Seven caries-free, intact, maxillary, and mandibular third molars from humans, aged 30-37 years, which were scheduled for extraction for orthodontic or surgical purposes, were included in the study. The patients received a thorough explanation of the experimental rationale, clinical procedures, and possible complications. All experimental protocols were independently reviewed and approved by the Local Ethics Committee of Pomeranian Medical University, Szczecin, Poland (approval number KB-0012/27/13).

Clinical protocol. For all included teeth, periapical radiographs were taken to exclude the presence of caries or periapical pathology. Tooth sensitivity was assessed by thermal testing (Kältespray; M&W Dental, Büdingen, Germany) and electric sensitivity testing (Vitality Scanner Pulp Vitality Tester; SybronEndo, Orange, CA, USA). These teeth were subjected to pulp exposure, direct capping with RetroMTA, and restoration with a composite resin. Seven months later, the teeth were clinically and radiographically evaluated. Clinical assessment was performed at 1 week and at 7 months after the procedure. During clinical interviews, the patients were asked about the presence of pain, and its type and duration. Reactions to thermal stimuli were classified into three categories: 1 = normal response (pain lasting up to 10 s); 2 = an extended response (pain > 10 s); 3 = no response. An electrical test was performed using a Vitality Scanner, and was repeated three times. Seven months after the procedure the teeth were extracted and subjected to histological processing and evaluation.

Histological processing. Immediately after extraction, the teeth were immersed in a 10% neutral buffered formalin solution, and gently washed from blood and saliva. After brief prefixation (≤10 minutes), special precautions were taken to facilitate pulp tissue fixation. The roots were separated 5 mm apically to the cemento-enamel junction, using a diamond disk under copious water cooling. Then the teeth were grinded with a high speed cylindrical diamond bur under water spray in a mesio-distal or bucco-lingual plane until exposing one or more pulp horns. Photographs and radiographs were taken of each sample before successive steps. For demineralization, the specimens were immersed for 3 to 4 weeks in an aqueous solution consisting of a mixture of 22.5% (v/v) formic acid and 10% (w/v) sodium citrate, with radiographic determination of the end-point. Then all specimens were washed in running tap water for 24 hours, dehydrated using ascending grades of ethanol, cleared in xylene, infiltrated, and embedded in paraffin (melting point of 56 °C) following standard procedures. The paraffin blocks were trimmed. With the microtome set at 5 μM, serial sections were taken until exhausting the entire pulp tissue in the chamber. Six to eight sections were collected on each slide. Every fifth slide was stained with haematoxylin and eosin for screening and evaluation of mineralized tissue formation. These stained sections were used to locate the areas exhibiting the most severe inflammatory reactions, and those with less favourable bridging. Based on this initial evaluation, all slides adjacent to the location with the less favourable conditions were stained. In addition, the selected slides were subjected to a modified Brown and Brenn technique (Taylor 1966) for staining bacteria. Next, cover slips were placed on the slides, and the sections were examined using a light microscope. For each pulp, the worst histologic condition observed was recorded. If bacteria were observed on the cavity walls or in the area of exposure, the case was excluded from evaluation.

Two intact teeth (one maxillary and one mandibular third molar) extracted for pericoronitis were used as control. To test the reliability of the bacterial stain, two teeth with deep caries were examined, extracted because deemed non-restorable. These teeth were processed using the same protocol as the experimental group.

Slides were observed under a light microscope (Leica DMLB; Leica Microsystems, Wetzlar, Germany) and digital photographs were taken (Leica DFC420; Leica Microsystems, Wetzlar, Germany). Following aspects were observed with particular care: 1) Presence and type of mineralized tissues formed in the area of the surgical exposure; 2) Morphology of cells layering this mineralized tissue; 3) Presence and degree of inflammatory reactions in the pulpal area subjacent to the newly formed tissue; and 4) Presence of stainable bacteria in the experimental cavity or the area of pulp exposure.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria were healthy patients with no contributing systemic conditions, who had at least one caries-free mature permanent third molar

Exclusion Criteria:

* The exclusion criteria included patients who had pulp inflammation, pulp necrosis, root resorption or periapical diseases

Ages: 30 Years to 37 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2016-04-03 (Actual); Primary Completion 2017-03-20 (Actual); Study Completion 2018-06-18 (Actual)

PRIMARY OUTCOMES:
Histological Evaluation of Direct Pulp Capping on Human Pulp Tissue Using a RetroMTA | 7 months
  Each histomorphologic section was scored from 1-3, with 1 representing the most desired result and 3 representing the least desired result.
  Mineralized tissue bridge
  1. Complete
  2. Incomplete
  3. Absent
  Mineralized tissue morphology
  1. Dentin associated with irregular hard tissue
  2. Only irregular hard tissue deposition
  3. No hard tissue deposition
  Inflammatory response
  1. Absent
  2. Mild (inflammatory cells next to dentin bridge or area of pulp exposure only)
  3. Severe (all of the coronal pulp is infiltrated or necrotic)
  Odontoblastic cell layer
  1. Presence of odontoblast cells and odontoblast-like cells
  2. Presence of odontoblast-like cells only
  3. Absent
  Presence of bacteria
  1. Absence
  2. Presence of stained bacterial profiles along the coronal or apical walls
  3. Presence of stained bacterial profiles within the dental pulp

SECONDARY OUTCOMES:
Clinical Examination of Direct Pulp Capping on Human Pulp Tissue Using a RetroMTA | 7 months
  Number of participants with adverse events related to RetroMTA treatment
  Periapical pathology
  1. absent
  2. present
  The presence of pain
  1. absent
  2. present
  Tooth sensitivity:
  I. Reactions to thermal stimuli
  1. present
  2. absent
  II. Electric sensitivity
  1. present
  2. absent
  1 representing the most desired result and 2 representing the least desired result.

CONTACTS AND LOCATIONS:
Overall Officials: Alicja Nowicka, DDS, PhD, Study Director — Department of Conservative Dentistry and Endodontics, Pomeranian Medical University, Al. Powstańców Wielkopolskich 72, 70-111, Szczecin, Poland; Till Dammaschke, DDS, PhD, Study Chair — Department of Periodontology and Operative Dentistry, Westphalian Wilhelms-University, Albert-Schweitzer-Campus 1, building W 30, 48149 Münster, Germany; Mariusz Lipski, DDS, PhD, Study Chair — Department of Preclinical Conservative Dentistry and Preclinical Endodontics, Pomeranian Medical University, Al. Powstańców Wielkopolskich 72, 70-111, Szczecin, Poland; Domenico Ricucci, MD, DDS, Study Chair — Private Practice, Piazza Calvario, 7, 87022 Cetraro (CS), Italy
Locations (1):
- Pomeranian Medical University in Szczecin, Szczecin, Rybacka 1, Poland

REFERENCES:
- [Derived] Dammaschke T, Nowicka A, Lipski M, Ricucci D. Histological evaluation of hard tissue formation after direct pulp capping with a fast-setting mineral trioxide aggregate (RetroMTA) in humans. Clin Oral Investig. 2019 Dec;23(12):4289-4299. doi: 10.1007/s00784-019-02876-2. Epub 2019 Mar 12. PMID 30864114